CLINICAL TRIAL: NCT02330419
Title: Better Than Study: Targeting Heavy Alcohol Use With Naltrexone Among MSM
Brief Title: Better Than Study: Targeting Heavy Alcohol Use With Naltrexone Among Men Who Have Sex With Men (MSM)
Acronym: SayWhen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco Department of Public Health (Other Government); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1DP5OD019809 (NIH); 1DP5OD019809 (NIH)
Record Dates: First submitted 2014-12-30; First posted 2015-01-05 (Estimated); Results first posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Binge Drinking; HIV
Keywords: Naltrexone
MeSH Terms: conditions — Binge Drinking | interventions — Naltrexone; Counseling; Ethanol; Urinalysis; Ecological Momentary Assessment

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo 50mg, as needed
  Interventions: Drug: Placebo; Behavioral: Medical Management (MM) counseling for alcohol use:; Diagnostic Test: Urinalysis for novel alcohol biochemical markers:; Behavioral: Behavioral survey measurements:; Diagnostic Test: Dried Blood Spot (DSB) Testing for Phosphatidylethanol; Behavioral: Ecological Momentary Assessment
- Naltrexone (Active Comparator): Naltrexone 50mg, as needed
  Interventions: Drug: Naltrexone; Behavioral: Medical Management (MM) counseling for alcohol use:; Diagnostic Test: Urinalysis for novel alcohol biochemical markers:; Behavioral: Behavioral survey measurements:; Diagnostic Test: Dried Blood Spot (DSB) Testing for Phosphatidylethanol; Behavioral: Ecological Momentary Assessment

INTERVENTIONS:
Drug: Placebo — Placebo capsules will contain microcrystalline cellulose (Medisca). Placebo and active medication will be provided in capsules that are an exact match in color, so as to make the placebo and active medication indistinguishable from each other.
  Arms: Placebo
Drug: Naltrexone — REVIA is a white, crystalline compound. The hydrochloride salt is soluble in water to the extent of about 100 mg/mL. REVIA is available in scored film-coated tablets containing 50 mg of naltrexone hydrochloride.
  Other Names: REVIA
  Arms: Naltrexone
Behavioral: Medical Management (MM) counseling for alcohol use: — MM is a low-intensity supportive program designed to increase problem recognition and enhance motivation to change maladaptive alcohol use patterns. Participants will receive individual 20 minute MM sessions weekly from trained staff supervised by a clinical psychologist
Diagnostic Test: Urinalysis for novel alcohol biochemical markers: — Urine samples will be collected weekly and tested for ethyl glucuronide (EtG) to determine recent alcohol consumption. EtG is a relatively novel, highly sensitive indicator for recent alcohol consumption; this alcohol biomarker is detectable in urine for approximately 72 hours).
  Other Names: Ethyl glucuronide
Behavioral: Behavioral survey measurements: — Standardized and validated behavioral measure that will be assessed using audio computer administered surveys (ACASI) to minimize underreporting of risk activities and standardize data collection
  Other Names: ACASI
Diagnostic Test: Dried Blood Spot (DSB) Testing for Phosphatidylethanol — Phosphatidylethanol (PEth)-a phospholipid formed only in the presence of alcohol-is a novel, direct biochemical marker of alcohol that has shown high (>95%) sensitivity and specificity to detect heavy drinking over a period of 2-3 weeks in several studies of dependent patients and abstainers. DSB samples will be collected at enrollment, weeks 3, 6, 9, 12, and post-treatment visits at month 1, 3, and 6.
Behavioral: Ecological Momentary Assessment — Ecological Momentary Assessments are SMS texts to collect data on alcohol consumption, number of drinks on drinking days, and targeted medication administration prior to anticipated drinking sessions. Messages will use short-hand notations to maintain participant confidentiality

SUMMARY:
This is a double-blind, placebo-controlled trial of 120 binge-drinking MSM to 12 weeks of naltrexone 50mg, to be taken in anticipation of heavy drinking. Ethnically and racially diverse participants will be recruited using Respondent Driven Sampling as well as active field recruitment. MSM will be seen weekly for alcohol-metabolite urine testing, study drug dispensing, and brief counseling for alcohol use. Safety assessments and behavioral surveys will be completed monthly.

DETAILED DESCRIPTION:
This is a double-blinded, placebo controlled trial of 120 binge-drinking MSM to 12 weeks of naltrexone 50mg, to be taken in anticipation of heavy drinking. Ethically and racially diverse participants will be recruited using venue based recruitment and social network bsed recruitment strategies. Participants will be seen weekly for alcohol metabolite urine testing, study drug dispensing and brief counseling for alcohol use. Safety assessments and behavioral surveys will be completed monthly. Efficacy on alcohol consumption and alcohol-associated sexual risk behavior (Aims 1-3) will be assessed using weekly timeline follow-back, screening for ethyl glucuronide (EtG) positive urines, and computer administered monthly interventions. Tolerability and acceptability (Aim 4) will be assessed through tracking of adverse events and medication adherence. Generalized estimating equation (GEE) models will be fitted to estimate treatment effects on repeated study outcomes.

ELIGIBILITY:
Inclusion Criteria:

* (1) Male gender (2) self-reported anal sex with men in the prior three months while under the influence of alcohol (3) at least one binge drinking (five or more drinks on a single occasion) session per week in the prior three months; (4) interested in reducing binge alcohol consumption; (5) HIV-negative by rapid antibody test or medical record documentation of HIV infection (HIV positive participants); (6) no current acute illnesses requiring prolonged medical care; (7) no chronic illnesses that are likely to progress clinically during trial participation; (8) able and willing to provide informed consent and adhere to visit schedule; (9) age 18-70 years; (10) baseline complete blood count (CBC), total protein, albumin, glucose, alkaline phosphatase, creatinine, blood urea nitrogen (BUN), and electrolytes without clinically significant abnormalities as determined by study clinician in conjunction with symptoms, physical exam, and medical history.

Exclusion Criteria:

* (1) Any psychiatric (e.g. depression with suicidal ideation) or medical condition that would preclude safe participation in the study; (2) known allergy/previous adverse reaction to naltrexone; (3) current use of/ dependence on any opioids or a known medical condition which currently requires/may likely require opioid analgesics; (4) opioid-positive urine at enrollment; (5) current CD4 count < 200 cells/mm3 (6) moderate/severe liver disease (aspartate aminotransferase (AST), alanine transaminase (ALT) > 3 times upper limit of normal); (7) impaired renal function (creatinine clearance < 50 ml/min); (8) currently participating in another intervention research study with potential overlap; (9) alcohol dependence as determined by Structured Clinical Interview for the Diagnostic and Statistical Manual for Mental Disorders (SCID) criteria (participants with non-dependent alcohol use disorders/symptoms of alcohol abuse (per Diagnostic and Statistical Manual--DSM-IV) are eligible) (10) any condition that, in the principal investigator and/or study clinician's judgment interferes with safe study participation or adherence to study procedures; (11) not having a cell-phone that can send and receive text messages.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn-Milo Santos, PhD, Principal Investigator — San Francisco Department of Public Health
Locations (1):
- Center on Substance Use and Health, San Francisco, California, United States

REFERENCES:
- [Background] Finlayson TJ, Le B, Smith A, Bowles K, Cribbin M, Miles I, Oster AM, Martin T, Edwards A, Dinenno E; Centers for Disease Control and Prevention (CDC). HIV risk, prevention, and testing behaviors among men who have sex with men--National HIV Behavioral Surveillance System, 21 U.S. cities, United States, 2008. MMWR Surveill Summ. 2011 Oct 28;60(14):1-34. PMID 22031280
- [Background] Centers for Disease Control and Prevention (CDC). Vital signs: binge drinking prevalence, frequency, and intensity among adults - United States, 2010. MMWR Morb Mortal Wkly Rep. 2012 Jan 13;61(1):14-9. PMID 22237031
- [Background] Stall R, Paul JP, Greenwood G, Pollack LM, Bein E, Crosby GM, Mills TC, Binson D, Coates TJ, Catania JA. Alcohol use, drug use and alcohol-related problems among men who have sex with men: the Urban Men's Health Study. Addiction. 2001 Nov;96(11):1589-601. doi: 10.1046/j.1360-0443.2001.961115896.x. PMID 11784456
- [Background] Colfax G, Vittinghoff E, Husnik MJ, McKirnan D, Buchbinder S, Koblin B, Celum C, Chesney M, Huang Y, Mayer K, Bozeman S, Judson FN, Bryant KJ, Coates TJ; EXPLORE Study Team. Substance use and sexual risk: a participant- and episode-level analysis among a cohort of men who have sex with men. Am J Epidemiol. 2004 May 15;159(10):1002-12. doi: 10.1093/aje/kwh135. PMID 15128613
- [Background] Wolitski RJ, Stall R, Valdiserri R. Unequal Opportunity: Health Disparities affecting Gay and Bisexual Men in the United States. New York: Oxford Press; 2008.
- [Background] Raymond HF. San Francisco National HIV Behavioral Surveillance Data - MSM and Binge-drinking. In: Santos GM, ed. San Francisco: San Francisco Department of Public Health; 2012.
- [Background] Raymond HF, Bereknyei S, Berglas N, Hunter J, Ojeda N, McFarland W. Estimating population size, HIV prevalence and HIV incidence among men who have sex with men: a case example of synthesising multiple empirical data sources and methods in San Francisco. Sex Transm Infect. 2013 Aug;89(5):383-7. doi: 10.1136/sextrans-2012-050675. Epub 2013 Apr 25. PMID 23620133
- [Background] Jin H. San Francisco National HIV Behavioral Surveillance Survey Data Request - MSM3 Binge Drinking Data. In: Santos G, ed. San Francisco2014:1.
- [Background] Prejean J, Song R, Hernandez A, Ziebell R, Green T, Walker F, Lin LS, An Q, Mermin J, Lansky A, Hall HI; HIV Incidence Surveillance Group. Estimated HIV incidence in the United States, 2006-2009. PLoS One. 2011;6(8):e17502. doi: 10.1371/journal.pone.0017502. Epub 2011 Aug 3. PMID 21826193
- [Background] SFDPH. HIV/AIDS Epidemiology Annual Report. San Francisco San Francisco Department of Public Health 2010.
- [Background] Mansergh G, Koblin BA, McKirnan DJ, Hudson SM, Flores SA, Wiegand RE, Purcell DW, Colfax GN; Project MIX Study Team. An intervention to reduce HIV risk behavior of substance-using men who have sex with men: a two-group randomized trial with a nonrandomized third group. PLoS Med. 2010 Aug 24;7(8):e1000329. doi: 10.1371/journal.pmed.1000329. PMID 20811491
- [Background] Leigh BC. Alcohol and condom use: a meta-analysis of event-level studies. Sex Transm Dis. 2002 Aug;29(8):476-82. doi: 10.1097/00007435-200208000-00008. PMID 12172533
- [Background] Woolf SE, Maisto SA. Alcohol use and risk of HIV infection among men who have sex with men. AIDS Behav. 2009 Aug;13(4):757-82. doi: 10.1007/s10461-007-9354-0. Epub 2008 Jan 31. PMID 18236149
- [Background] Maisto SA, Palfai T, Vanable PA, Heath J, Woolf-King SE. The effects of alcohol and sexual arousal on determinants of sexual risk in men who have sex with men. Arch Sex Behav. 2012 Aug;41(4):971-86. doi: 10.1007/s10508-011-9846-x. Epub 2011 Oct 19. PMID 22009480
- [Background] George WH, Stoner SA. Understanding acute alcohol effects on sexual behavior. Annu Rev Sex Res. 2000;11:92-124. PMID 11351836
- [Background] Howard J, Taylor JA, Ganikos ML, Holder HD, Godwin DF, Taylor ED. An overview of prevention research: issues, answers, and new agendas. Public Health Rep. 1988 Nov-Dec;103(6):674-83. PMID 3141964
- [Background] Cooper ML. Alcohol use and risky sexual behavior among college students and youth: evaluating the evidence. J Stud Alcohol Suppl. 2002 Mar;(14):101-17. doi: 10.15288/jsas.2002.s14.101. PMID 12022716
- [Background] George WH, Stoner SA, Norris J, Lopez PA, Lehman GL. Alcohol expectancies and sexuality: a self-fulfilling prophecy analysis of dyadic perceptions and behavior. J Stud Alcohol. 2000 Jan;61(1):168-76. doi: 10.15288/jsa.2000.61.168. PMID 10627112
- [Background] Steele CM, Josephs RA. Alcohol myopia. Its prized and dangerous effects. Am Psychol. 1990 Aug;45(8):921-33. doi: 10.1037//0003-066x.45.8.921. PMID 2221564
- [Background] McKirnan DJ, Ostrow DG, Hope B. Sex, drugs and escape: a psychological model of HIV-risk sexual behaviours. AIDS Care. 1996 Dec;8(6):655-69. doi: 10.1080/09540129650125371. PMID 8993716
- [Background] Heatherton TF, Baumeister RF. Binge eating as escape from self-awareness. Psychol Bull. 1991 Jul;110(1):86-108. doi: 10.1037/0033-2909.110.1.86. PMID 1891520
- [Background] Cooper ML, Orcutt HK. Alcohol use, condom use and partner type among heterosexual adolescents and young adults. J Stud Alcohol. 2000 May;61(3):413-9. doi: 10.15288/jsa.2000.61.413. PMID 10807212
- [Background] Leigh BC, Stacy AW. Alcohol expectancies and drinking in different age groups. Addiction. 2004 Feb;99(2):215-27. doi: 10.1111/j.1360-0443.2003.00641.x. PMID 14756714
- [Background] Stueve A, O'Donnell L, Duran R, San Doval A, Geier J; Community Intervention Trial for Youth Study Team. Being high and taking sexual risks: findings from a multisite survey of urban young men who have sex with men. AIDS Educ Prev. 2002 Dec;14(6):482-95. doi: 10.1521/aeap.14.8.482.24108. PMID 12512849
- [Background] Fergus S, Lewis MA, Darbes LA, Butterfield RM. HIV risk and protection among gay male couples: the role of gay community integration. Health Educ Behav. 2005 Apr;32(2):151-71. doi: 10.1177/1090198104271964. PMID 15856614
- [Background] Voetsch AC, Lansky A, Drake AJ, MacKellar D, Bingham TA, Oster AM, Sullivan PS. Comparison of demographic and behavioral characteristics of men who have sex with men by enrollment venue type in the National HIV Behavioral Surveillance System. Sex Transm Dis. 2012 Mar;39(3):229-35. doi: 10.1097/OLQ.0b013e31823d2b24. PMID 22337112
- [Background] Vosburgh HW, Mansergh G, Sullivan PS, Purcell DW. A review of the literature on event-level substance use and sexual risk behavior among men who have sex with men. AIDS Behav. 2012 Aug;16(6):1394-410. doi: 10.1007/s10461-011-0131-8. PMID 22323004
- [Background] Vanable PA, McKirnan DJ, Buchbinder SP, Bartholow BN, Douglas JM Jr, Judson FN, MacQueen KM. Alcohol use and high-risk sexual behavior among men who have sex with men: the effects of consumption level and partner type. Health Psychol. 2004 Sep;23(5):525-32. doi: 10.1037/0278-6133.23.5.525. PMID 15367072
- [Background] Irwin TW, Morgenstern J, Parsons JT, Wainberg M, Labouvie E. Alcohol and sexual HIV risk behavior among problem drinking men who have sex with men: An event level analysis of timeline followback data. AIDS Behav. 2006 May;10(3):299-307. doi: 10.1007/s10461-005-9045-7. PMID 16482407
- [Background] Prestage G, Grierson J, Bradley J, Hurley M, Hudson J. The role of drugs during group sex among gay men in Australia. Sex Health. 2009 Dec;6(4):310-7. doi: 10.1071/SH09014. PMID 19917200
- [Background] Benotsch EG, Nettles CD, Wong F, Redmann J, Boschini J, Pinkerton SD, Ragsdale K, Mikytuck JJ. Sexual risk behavior in men attending Mardi Gras celebrations in New Orleans, Louisiana. J Community Health. 2007 Oct;32(5):343-56. doi: 10.1007/s10900-007-9054-8. PMID 17922205
- [Background] Benotsch EG, Mikytuck JJ, Ragsdale K, Pinkerton SD. Sexual risk and HIV acquisition among men who have sex with men travelers to Key West, Florida: a mathematical modeling analysis. AIDS Patient Care STDS. 2006 Aug;20(8):549-56. doi: 10.1089/apc.2006.20.549. PMID 16893324
- [Background] Lambert G, Cox J, Hottes TS, Tremblay C, Frigault LR, Alary M, Otis J, Remis RS; M-Track Study Group. Correlates of unprotected anal sex at last sexual episode: analysis from a surveillance study of men who have sex with men in Montreal. AIDS Behav. 2011 Apr;15(3):584-95. doi: 10.1007/s10461-009-9605-3. PMID 20033763
- [Background] Folch C, Esteve A, Zaragoza K, Munoz R, Casabona J. Correlates of intensive alcohol and drug use in men who have sex with men in Catalonia, Spain. Eur J Public Health. 2010 Apr;20(2):139-45. doi: 10.1093/eurpub/ckp091. Epub 2009 Jun 29. PMID 19564240
- [Background] Reisner SL, Mimiaga MJ, Case P, Johnson CV, Safren SA, Mayer KH. Predictors of identifying as a barebacker among high-risk New England HIV seronegative men who have sex with men. J Urban Health. 2009 Mar;86(2):250-62. doi: 10.1007/s11524-008-9333-4. Epub 2008 Dec 3. PMID 19051039
- [Background] NYCDOHMH. Alcohol use and risky sex in New York City. New York City: New York City Department of Health and Mental Hygiene;2008.
- [Background] Mackesy-Amiti ME, Fendrich M, Johnson TP. Symptoms of substance dependence and risky sexual behavior in a probability sample of HIV-negative men who have sex with men in Chicago. Drug Alcohol Depend. 2010 Jul 1;110(1-2):38-43. doi: 10.1016/j.drugalcdep.2010.01.016. Epub 2010 Mar 9. PMID 20219291
- [Background] Reisner SL, Mimiaga MJ, Bland S, Skeer M, Cranston K, Isenberg D, Driscoll M, Mayer KH. Problematic alcohol use and HIV risk among Black men who have sex with men in Massachusetts. AIDS Care. 2010 May;22(5):577-87. doi: 10.1080/09540120903311482. PMID 20336557
- [Background] Mimiaga MJ, Thomas B, Mayer KH, Reisner SL, Menon S, Swaminathan S, Periyasamy M, Johnson CV, Safren SA. Alcohol use and HIV sexual risk among MSM in Chennai, India. Int J STD AIDS. 2011 Mar;22(3):121-5. doi: 10.1258/ijsa.2009.009059. PMID 21464447
- [Background] Nelson KM, Simoni JM, Pearson CR, Walters KL. 'I've had unsafe sex so many times why bother being safe now?': the role of cognitions in sexual risk among American Indian/Alaska Native men who have sex with men. Ann Behav Med. 2011 Dec;42(3):370-80. doi: 10.1007/s12160-011-9302-0. PMID 21887585
- [Background] Read TR, Hocking J, Sinnott V, Hellard M. Risk factors for incident HIV infection in men having sex with men: a case-control study. Sex Health. 2007 Mar;4(1):35-9. doi: 10.1071/sh06043. PMID 17382036
- [Background] Koblin BA, Husnik MJ, Colfax G, Huang Y, Madison M, Mayer K, Barresi PJ, Coates TJ, Chesney MA, Buchbinder S. Risk factors for HIV infection among men who have sex with men. AIDS. 2006 Mar 21;20(5):731-9. doi: 10.1097/01.aids.0000216374.61442.55. PMID 16514304
- [Background] Sander PM, Cole SR, Stall RD, Jacobson LP, Eron JJ, Napravnik S, Gaynes BN, Johnson-Hill LM, Bolan RK, Ostrow DG. Joint effects of alcohol consumption and high-risk sexual behavior on HIV seroconversion among men who have sex with men. AIDS. 2013 Mar 13;27(5):815-23. doi: 10.1097/QAD.0b013e32835cff4b. PMID 23719351
- [Background] Santos GM, Das M, Colfax GN. Interventions for non-injection substance use among US men who have sex with men: what is needed. AIDS Behav. 2011 Apr;15 Suppl 1(Suppl 1):S51-6. doi: 10.1007/s10461-011-9923-0. No abstract available. PMID 21404011
- [Background] Paul JP, Barrett DC, Crosby GM, Stall RD. Longitudinal changes in alcohol and drug use among men seen at a gay-specific substance abuse treatment agency. J Stud Alcohol. 1996 Sep;57(5):475-85. doi: 10.15288/jsa.1996.57.475. PMID 8858545
- [Background] Fals-Stewart W, O'Farrell TJ, Lam WK. Behavioral couple therapy for gay and lesbian couples with alcohol use disorders. J Subst Abuse Treat. 2009 Dec;37(4):379-87. doi: 10.1016/j.jsat.2009.05.001. Epub 2009 Jun 23. PMID 19553063
- [Background] Bux D. The epidemiology of problem drinking in gay men and lesbians: A Critical Review. Clinical Psychology Review. 1996;16(4):277-298.
- [Background] Colfax GN, Santos GM, Das M, Santos DM, Matheson T, Gasper J, Shoptaw S, Vittinghoff E. Mirtazapine to reduce methamphetamine use: a randomized controlled trial. Arch Gen Psychiatry. 2011 Nov;68(11):1168-75. doi: 10.1001/archgenpsychiatry.2011.124. PMID 22065532
- [Background] Shoptaw S, Reback CJ, Frosch DL, Rawson RA. Stimulant abuse treatment as HIV prevention. J Addict Dis. 1998;17(4):19-32. doi: 10.1300/J069v17n04_03. PMID 9848029
- [Background] Ulm RR, Volpicelli JR, Volpicelli LA. Opiates and alcohol self-administration in animals. J Clin Psychiatry. 1995;56 Suppl 7:5-14. PMID 7673105
- [Background] Ray LA, Chin PF, Miotto K. Naltrexone for the treatment of alcoholism: clinical findings, mechanisms of action, and pharmacogenetics. CNS Neurol Disord Drug Targets. 2010 Mar;9(1):13-22. doi: 10.2174/187152710790966704. PMID 20201811
- [Background] Alkermes. Vivitrol - Mechanism of action for alcohol dependence. http://www.vivitrol.com/hcptreating/howvivitrolworks. Published 2012. Accessed 03/01/2012.
- [Background] Magendzo K, Bustos G. Expression of amphetamine-induced behavioral sensitization after short- and long-term withdrawal periods: participation of mu- and delta-opioid receptors. Neuropsychopharmacology. 2003 Mar;28(3):468-77. doi: 10.1038/sj.npp.1300063. Epub 2002 Sep 13. PMID 12629526
- [Background] Chiu CT, Ma T, Ho IK. Methamphetamine-induced behavioral sensitization in mice: alterations in mu-opioid receptor. J Biomed Sci. 2006 Nov;13(6):797-811. doi: 10.1007/s11373-006-9102-x. Epub 2006 Jul 18. PMID 16847721
- [Background] Schad CA, Justice JB Jr, Holtzman SG. Endogenous opioids in dopaminergic cell body regions modulate amphetamine-induced increases in extracellular dopamine levels in the terminal regions. J Pharmacol Exp Ther. 2002 Mar;300(3):932-8. doi: 10.1124/jpet.300.3.932. PMID 11861800
- [Background] Trujillo KA, Belluzzi JD, Stein L. Naloxone blockade of amphetamine place preference conditioning. Psychopharmacology (Berl). 1991;104(2):265-74. doi: 10.1007/BF02244190. PMID 1876671
- [Background] Altshuler HL, Phillips PE, Feinhandler DA. Alteration of ethanol self-administration by naltrexone. Life Sci. 1980 Mar 3;26(9):679-88. doi: 10.1016/0024-3205(80)90257-x. No abstract available. PMID 6767889
- [Background] Volpicelli JR, Watson NT, King AC, Sherman CE, O'Brien CP. Effect of naltrexone on alcohol "high" in alcoholics. Am J Psychiatry. 1995 Apr;152(4):613-5. doi: 10.1176/ajp.152.4.613. PMID 7694913
- [Background] Batki SL, Dimmock JA, Ploutz-Snyder R, Meszaros ZS, Canfield K. Directly Monitored Naltrexone Reduces Heavy Drinking in Schizophrenia: Preliminary Analysis of a Controlled Trial. Alcoholism Clinical and Experimental Research. 2009;33(6):116A.
- [Background] Batki SL, Dimmock JA, Wade M, Gately PW, Cornell M, Maisto SA, Carey KB, Ploutz-Snyder R. Monitored naltrexone without counseling for alcohol abuse/dependence in schizophrenia-spectrum disorders. Am J Addict. 2007 Jul-Aug;16(4):253-9. doi: 10.1080/10550490701389732. PMID 17661192
- [Background] King AC, de Wit H, McNamara PJ, Cao D. Rewarding, stimulant, and sedative alcohol responses and relationship to future binge drinking. Arch Gen Psychiatry. 2011 Apr;68(4):389-99. doi: 10.1001/archgenpsychiatry.2011.26. PMID 21464363
- [Background] O'Malley SS, Jaffe AJ, Chang G, Schottenfeld RS, Meyer RE, Rounsaville B. Naltrexone and coping skills therapy for alcohol dependence. A controlled study. Arch Gen Psychiatry. 1992 Nov;49(11):881-7. doi: 10.1001/archpsyc.1992.01820110045007. PMID 1444726
- [Background] Volpicelli JR, Rhines KC, Rhines JS, Volpicelli LA, Alterman AI, O'Brien CP. Naltrexone and alcohol dependence. Role of subject compliance. Arch Gen Psychiatry. 1997 Aug;54(8):737-42. doi: 10.1001/archpsyc.1997.01830200071010. PMID 9283509
- [Background] Chick J, Anton R, Checinski K, Croop R, Drummond DC, Farmer R, Labriola D, Marshall J, Moncrieff J, Morgan MY, Peters T, Ritson B. A multicentre, randomized, double-blind, placebo-controlled trial of naltrexone in the treatment of alcohol dependence or abuse. Alcohol Alcohol. 2000 Nov-Dec;35(6):587-93. doi: 10.1093/alcalc/35.6.587. PMID 11093966
- [Background] Croop RS, Faulkner EB, Labriola DF. The safety profile of naltrexone in the treatment of alcoholism. Results from a multicenter usage study. The Naltrexone Usage Study Group. Arch Gen Psychiatry. 1997 Dec;54(12):1130-5. doi: 10.1001/archpsyc.1997.01830240090013. PMID 9400350
- [Background] Prescribing Information Naltrexone Hydrochloride Tablets USP. Mallinckrodt Inc. http://pharmaceuticals.mallinckrodt.com/_attachments/PackageInserts/35_Naltrexone%20HCl%20Tablets_REV020509.pdf. Published 2009. Accessed April 22, 2010, 2010.
- [Background] Anton RF, O'Malley SS, Ciraulo DA, Cisler RA, Couper D, Donovan DM, Gastfriend DR, Hosking JD, Johnson BA, LoCastro JS, Longabaugh R, Mason BJ, Mattson ME, Miller WR, Pettinati HM, Randall CL, Swift R, Weiss RD, Williams LD, Zweben A; COMBINE Study Research Group. Combined pharmacotherapies and behavioral interventions for alcohol dependence: the COMBINE study: a randomized controlled trial. JAMA. 2006 May 3;295(17):2003-17. doi: 10.1001/jama.295.17.2003. PMID 16670409
- [Background] Brewer C, Wong VS. Naltrexone: report of lack of hepatotoxicity in acute viral hepatitis, with a review of the literature. Addict Biol. 2004 Mar;9(1):81-7. doi: 10.1080/13556210410001674130. PMID 15203443
- [Background] Monti PM, Rohsenow DJ, Swift RM, Gulliver SB, Colby SM, Mueller TI, Brown RA, Gordon A, Abrams DB, Niaura RS, Asher MK. Naltrexone and cue exposure with coping and communication skills training for alcoholics: treatment process and 1-year outcomes. Alcohol Clin Exp Res. 2001 Nov;25(11):1634-47. PMID 11707638
- [Background] Lee MC, Wagner HN Jr, Tanada S, Frost JJ, Bice AN, Dannals RF. Duration of occupancy of opiate receptors by naltrexone. J Nucl Med. 1988 Jul;29(7):1207-11. PMID 2839637
- [Background] Leeman RF, Palmer RS, Corbin WR, Romano DM, Meandzija B, O'Malley SS. A pilot study of naltrexone and BASICS for heavy drinking young adults. Addict Behav. 2008 Aug;33(8):1048-54. doi: 10.1016/j.addbeh.2008.04.007. Epub 2008 Apr 13. PMID 18502591
- [Background] Kranzler HR, Armeli S, Feinn R, Tennen H. Targeted naltrexone treatment moderates the relations between mood and drinking behavior among problem drinkers. J Consult Clin Psychol. 2004 Apr;72(2):317-27. doi: 10.1037/0022-006X.72.2.317. PMID 15065964
- [Background] Kranzler HR, Armeli S, Tennen H, Blomqvist O, Oncken C, Petry N, Feinn R. Targeted naltrexone for early problem drinkers. J Clin Psychopharmacol. 2003 Jun;23(3):294-304. doi: 10.1097/01.jcp.0000084030.22282.6d. PMID 12826991
- [Background] Kranzler HR, Tennen H, Armeli S, Chan G, Covault J, Arias A, Oncken C. Targeted naltrexone for problem drinkers. J Clin Psychopharmacol. 2009 Aug;29(4):350-7. doi: 10.1097/JCP.0b013e3181ac5213. PMID 19593174
- [Background] Kranzler HR, Tennen H, Penta C, Bohn MJ. Targeted naltrexone treatment of early problem drinkers. Addict Behav. 1997 May-Jun;22(3):431-6. doi: 10.1016/s0306-4603(96)00064-0. PMID 9183513
- [Background] Heinala P, Alho H, Kiianmaa K, Lonnqvist J, Kuoppasalmi K, Sinclair JD. Targeted use of naltrexone without prior detoxification in the treatment of alcohol dependence: a factorial double-blind, placebo-controlled trial. J Clin Psychopharmacol. 2001 Jun;21(3):287-92. doi: 10.1097/00004714-200106000-00006. PMID 11386491
- [Background] Karhuvaara S, Simojoki K, Virta A, Rosberg M, Loyttyniemi E, Nurminen T, Kallio A, Makela R. Targeted nalmefene with simple medical management in the treatment of heavy drinkers: a randomized double-blind placebo-controlled multicenter study. Alcohol Clin Exp Res. 2007 Jul;31(7):1179-87. doi: 10.1111/j.1530-0277.2007.00401.x. Epub 2007 Apr 19. PMID 17451401
- [Background] Trial watch: Nalmefene reduces alcohol use in phase III trial. Nat Rev Drug Discov. 2011 Aug 1;10(8):566. doi: 10.1038/nrd3518. No abstract available. PMID 21804585
- [Background] Batki SL, Dimmock JA, Meszaros ZS, et al. Extended-Release Naltrexone for Alcohol Dependence in Serious Mental Illness. Alcoholism Clinical and Experimental Research
- [Background] Das M, Santos D, Matheson T, Santos GM, Chu P, Vittinghoff E, Shoptaw S, Colfax GN. Feasibility and acceptability of a phase II randomized pharmacologic intervention for methamphetamine dependence in high-risk men who have sex with men. AIDS. 2010 Apr 24;24(7):991-1000. doi: 10.1097/qad.0b013e328336e98b. PMID 20397286
- [Background] Coffin PO, Santos GM, Das M, Santos DM, Huffaker S, Matheson T, Gasper J, Vittinghoff E, Colfax GN. Aripiprazole for the treatment of methamphetamine dependence: a randomized, double-blind, placebo-controlled trial. Addiction. 2013 Apr;108(4):751-61. doi: 10.1111/add.12073. Epub 2013 Jan 3. PMID 23186131
- [Background] Coffin PO, Santos GM, Colfax G, Das M, Matheson T, DeMicco E, Dilley J, Vittinghoff E, Raiford JL, Carry M, Herbst JH. Adapted personalized cognitive counseling for episodic substance-using men who have sex with men: a randomized controlled trial. AIDS Behav. 2014 Jul;18(7):1390-400. doi: 10.1007/s10461-014-0712-4. PMID 24510401
- [Background] Das M, Dadasovich R, Matheson T, et al. Adapting an Effective HIV Prevention Intervention, Personalized Cognitive Counseling, for Episodic Substance-Using Men who have Sex with Men (SUMSM). XVIII International AIDS Conference; 07/14/2010, 2010; Vienna, Austria. Abstract #WEPE0324
- [Background] Colfax G, Santos GM, Chu P, Vittinghoff E, Pluddemann A, Kumar S, Hart C. Amphetamine-group substances and HIV. Lancet. 2010 Aug 7;376(9739):458-74. doi: 10.1016/S0140-6736(10)60753-2. PMID 20650520
- [Background] Santos GM, Das M, Santos D, Chu P, Vittinghoff E, G. C. Adherence in pharmacotherapy trials among methamphetamine-dependent men who have sex with men (MSM). . North American Congress of Epidemiology. Abstract# 00003039 June, 2011 2011; Montreal, QC
- [Background] Santos GM, Das M, Matheson T, Vittinghoff E, Dilley J, Colfax G. High-risk sexual behaviors associated with increasing combinations of polysubstances among substance-using men who have sex with men (SUMSM). Abstract# A-452-0270-13751. XIX International AIDS Conference (AIDS 2012). ; July, 2012, 2012; Washington, D.C.
- [Background] Santos GM, Das M, Santos D, Chu P, G. C. Social network analysis of methamphetamine-using men who have sex with men in San Francisco. 2011 National HIV Prevention Conference. Abstract# 1463 August, 2011., 2011; Atlanta, GA.
- [Background] Santos GM, Do T, Beck J, Makofane K, Arreola S, Pyun T, Hebert P, Wilson PA, Ayala G. Syndemic conditions associated with increased HIV risk in a global sample of men who have sex with men. Sex Transm Infect. 2014 May;90(3):250-3. doi: 10.1136/sextrans-2013-051318. Epub 2014 Jan 15. PMID 24431183
- [Background] Santos GM, Beck J, Wilson PA, Hebert P, Makofane K, Pyun T, Do T, Arreola S, Ayala G. Homophobia as a barrier to HIV prevention service access for young men who have sex with men. J Acquir Immune Defic Syndr. 2013 Aug 15;63(5):e167-70. doi: 10.1097/QAI.0b013e318294de80. No abstract available. PMID 24135782
- [Background] Silva-Santisteban A, Raymond HF, Salazar X, Villayzan J, Leon S, McFarland W, Caceres CF. Understanding the HIV/AIDS epidemic in transgender women of Lima, Peru: results from a sero-epidemiologic study using respondent driven sampling. AIDS Behav. 2012 May;16(4):872-81. doi: 10.1007/s10461-011-0053-5. PMID 21983694
- [Background] Ruan S, Yang H, Zhu Y, Ma Y, Li J, Zhao J, McFarland W, Raymond HF. HIV prevalence and correlates of unprotected anal intercourse among men who have sex with men, Jinan, China. AIDS Behav. 2008 May;12(3):469-75. doi: 10.1007/s10461-008-9361-9. Epub 2008 Feb 8. PMID 18259850
- [Background] Malekinejad M, McFarland W, Vaudrey J, Raymond HF. Accessing a diverse sample of injection drug users in San Francisco through respondent-driven sampling. Drug Alcohol Depend. 2011 Nov 1;118(2-3):83-91. doi: 10.1016/j.drugalcdep.2011.03.002. Epub 2011 Mar 24. PMID 21435803
- [Background] Lane T, Raymond HF, Dladla S, Rasethe J, Struthers H, McFarland W, McIntyre J. High HIV prevalence among men who have sex with men in Soweto, South Africa: results from the Soweto Men's Study. AIDS Behav. 2011 Apr;15(3):626-34. doi: 10.1007/s10461-009-9598-y. Epub 2009 Aug 7. PMID 19662523
- [Background] Raymond HF, Kajubi P, Kamya MR, Rutherford GW, Mandel JS, McFarland W. Correlates of unprotected receptive anal intercourse among gay and bisexual men: Kampala, Uganda. AIDS Behav. 2009 Aug;13(4):677-81. doi: 10.1007/s10461-009-9557-7. Epub 2009 Jun 3. PMID 19495955
- [Background] Jenkins RA. Recruiting substance-using men who have sex with men into HIV prevention research: current status and future directions. AIDS Behav. 2012 Aug;16(6):1411-9. doi: 10.1007/s10461-011-0037-5. PMID 22016329
- [Background] Heckathorn DD. Extensions of responder-driven sampling: analyzing continuous variables and controlling for differential recruitment. Sociol Methodol. 2007;37:151-207.
- [Background] Magnani R, Sabin K, Saidel T, Heckathorn D. Review of sampling hard-to-reach and hidden populations for HIV surveillance. AIDS. 2005 May;19 Suppl 2:S67-72. doi: 10.1097/01.aids.0000172879.20628.e1. PMID 15930843
- [Background] Wejnert C, Heckathorn DD. Web-Based Network Sampling. Sociological Methods & Research. 2008;37(1):105-134.
- [Background] McKnight C, Des Jarlais D, Bramson H, Tower L, Abdul-Quader AS, Nemeth C, Heckathorn D. Respondent-driven sampling in a study of drug users in New York City: notes from the field. J Urban Health. 2006 Nov;83(6 Suppl):i54-9. doi: 10.1007/s11524-006-9102-1. PMID 16977493
- [Background] Kamb ML, Fishbein M, Douglas JM Jr, Rhodes F, Rogers J, Bolan G, Zenilman J, Hoxworth T, Malotte CK, Iatesta M, Kent C, Lentz A, Graziano S, Byers RH, Peterman TA. Efficacy of risk-reduction counseling to prevent human immunodeficiency virus and sexually transmitted diseases: a randomized controlled trial. Project RESPECT Study Group. JAMA. 1998 Oct 7;280(13):1161-7. doi: 10.1001/jama.280.13.1161. PMID 9777816
- [Background] Pettinati HM, Weiss R, Miller WR, Donovan D, Ernst DB, Rounsaville BJ. Medical Management Treatment Manual: A Clinical Research Guide for Medically Trained Clinicians Providing Pharmacotherapy as Part of the Treatment for Alcohol Dependence. . Bethesda, MD: NIAAA;2004.
- [Background] Koblin B, Chesney M, Coates T; EXPLORE Study Team. Effects of a behavioural intervention to reduce acquisition of HIV infection among men who have sex with men: the EXPLORE randomised controlled study. Lancet. 2004 Jul 3-9;364(9428):41-50. doi: 10.1016/S0140-6736(04)16588-4. PMID 15234855
- [Background] Macalino GE, Celentano DD, Latkin C, Strathdee SA, Vlahov D. Risk behaviors by audio computer-assisted self-interviews among HIV-seropositive and HIV-seronegative injection drug users. AIDS Educ Prev. 2002 Oct;14(5):367-78. doi: 10.1521/aeap.14.6.367.24075. PMID 12413183
- [Background] Sobell L, Sobell M. Timeline follow-back: a technique for assessing self-reported alcohol consumption. In: Litten R, Allen J, eds. Measuring Alcohol Consumption. New York: Humana Press; 1992:41-72.
- [Background] Koblin BA, Chesney MA, Husnik MJ, Bozeman S, Celum CL, Buchbinder S, Mayer K, McKirnan D, Judson FN, Huang Y, Coates TJ; EXPLORE Study Team. High-risk behaviors among men who have sex with men in 6 US cities: baseline data from the EXPLORE Study. Am J Public Health. 2003 Jun;93(6):926-32. doi: 10.2105/ajph.93.6.926. PMID 12773357
- [Background] DAIDS. Table for grading severity of adult adverse experiences for prevention research programs. http://www.hptn.org/Web%20Documents/Regulatory_Resources/VPRP_toxtables.pdf. Published 2003. Accessed December, 2004.
- [Background] Maisto SA, Saitz R. Alcohol use disorders: screening and diagnosis. Am J Addict. 2003;12(s1):s12-s25. doi: 10.1111/j.1521-0391.2003.tb00493.x. PMID 14972777
- [Background] Cheng ST, Chan AC, Fung HH. Factorial structure of a short version of the Center for Epidemiologic Studies Depression Scale. Int J Geriatr Psychiatry. 2006 Apr;21(4):333-6. doi: 10.1002/gps.1467. PMID 16570325
- [Background] Derogatis LR, Melisaratos N. The Brief Symptom Inventory: an introductory report. Psychol Med. 1983 Aug;13(3):595-605. PMID 6622612
- [Background] Gossop M, Darke S, Griffiths P, Hando J, Powis B, Hall W, Strang J. The Severity of Dependence Scale (SDS): psychometric properties of the SDS in English and Australian samples of heroin, cocaine and amphetamine users. Addiction. 1995 May;90(5):607-14. doi: 10.1046/j.1360-0443.1995.9056072.x. PMID 7795497
- [Background] Han DH, Bolo N, Daniels MA, Lyoo IK, Min KJ, Kim CH, Renshaw PF. Craving for alcohol and food during treatment for alcohol dependence: modulation by T allele of 1519T>C GABAAalpha6. Alcohol Clin Exp Res. 2008 Sep;32(9):1593-9. doi: 10.1111/j.1530-0277.2008.00734.x. Epub 2008 Jul 9. PMID 18616664
- [Background] DAIDS. Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events In:2009.
- [Background] Haberer JE, Kahane J, Kigozi I, Emenyonu N, Hunt P, Martin J, Bangsberg DR. Real-time adherence monitoring for HIV antiretroviral therapy. AIDS Behav. 2010 Dec;14(6):1340-6. doi: 10.1007/s10461-010-9799-4. PMID 20809380
- [Background] Litten RZ, Bradley AM, Moss HB. Alcohol biomarkers in applied settings: recent advances and future research opportunities. Alcohol Clin Exp Res. 2010 Jun;34(6):955-67. doi: 10.1111/j.1530-0277.2010.01170.x. Epub 2010 Apr 5. PMID 20374219
- [Background] SAMHSA. The Role of Biomarkers in the Treatment of Alcohol Use Disorders, 2012 Revision. SAMHSA Advisory. 2012;11(2):1-8
- [Background] Kalapatapu RK, Chambers R. Novel Objective Biomarkers of Alcohol Use: Potential Diagnostic and Treatment Management Tools in Dual Diagnosis Care. J Dual Diagn. 2009 Jan 1;5(1):57-82. doi: 10.1080/15504260802628684. PMID 20582236
- [Background] Jatlow P, O'Malley SS. Clinical (nonforensic) application of ethyl glucuronide measurement: are we ready? Alcohol Clin Exp Res. 2010 Jun;34(6):968-75. doi: 10.1111/j.1530-0277.2010.01171.x. Epub 2010 Apr 5. PMID 20374218
- [Background] Santos GM, Lasher BA, Heinz AJ, et al. Urinary Ethyl Glucuronide and Ethyl Sulfate Testing to Evaluate the Efficacy of Topiramate for Alcohol Dependence Among Veterans with Post-Traumatic Stress Disorder. Research Society on Alcoholism; June 22, 2013, 2013; Orlando, FL.
- [Background] Laird NM. Missing data in longitudinal studies. Stat Med. 1988 Jan-Feb;7(1-2):305-15. doi: 10.1002/sim.4780070131. PMID 3353609
- [Background] Little RJA. Modeling the drop-out mechanism in repeated-measures studies. J Amer Stat Assoc. 1995;90(431):1112-1121.
- [Background] Robins JM, Rotnizky A, Zhao LP. Analysis of semiparametric regression models for repeated outcomes in the presence of missing data. J Amer Stat Assoc. 1995;90(429):106-121.
- [Background] Hartz DT, Frederick-Osborne SL, Galloway GP. Craving predicts use during treatment for methamphetamine dependence: a prospective, repeated-measures, within-subject analysis. Drug Alcohol Depend. 2001 Aug 1;63(3):269-76. doi: 10.1016/s0376-8716(00)00217-9. PMID 11418231
- [Background] Cole SR, Hernan MA. Fallibility in estimating direct effects. Int J Epidemiol. 2002 Feb;31(1):163-5. doi: 10.1093/ije/31.1.163. PMID 11914314
- [Background] Robins JM, Hernan MA, Brumback B. Marginal structural models and causal inference in epidemiology. Epidemiology. 2000 Sep;11(5):550-60. doi: 10.1097/00001648-200009000-00011. PMID 10955408
- [Background] Hernan MA, Brumback B, Robins JM. Marginal structural models to estimate the joint causal effect of nonrandomized treatments. J Amer Stat Assoc. 2001;96(454):440-448
- [Background] Jayaram-Lindstrom N, Hammarberg A, Beck O, Franck J. Naltrexone for the treatment of amphetamine dependence: a randomized, placebo-controlled trial. Am J Psychiatry. 2008 Nov;165(11):1442-8. doi: 10.1176/appi.ajp.2008.08020304. Epub 2008 Sep 2. PMID 18765480
- [Background] Jayaram-Lindstrom N, Konstenius M, Eksborg S, Beck O, Hammarberg A, Franck J. Naltrexone attenuates the subjective effects of amphetamine in patients with amphetamine dependence. Neuropsychopharmacology. 2008 Jul;33(8):1856-63. doi: 10.1038/sj.npp.1301572. Epub 2007 Oct 24. PMID 17957221
- [Background] Roozen HG, de Waart R, van den Brink W. Efficacy and tolerability of naltrexone in the treatment of alcohol dependence: oral versus injectable delivery. Eur Addict Res. 2007;13(4):201-6. doi: 10.1159/000104882. PMID 17851241
- [Background] FDA U. Naltrexone for extended-release injectable suspension (marketed as Vivitrol) information. http://www.fda.gov/Drugs/DrugSafety/PostmarketDrugSafetyInformationforPatientsandProviders/ucm103334.htm. Published 2008. Accessed April 27. 2010, 2010.
- [Background] Heilig M, Egli M. Pharmacological treatment of alcohol dependence: target symptoms and target mechanisms. Pharmacol Ther. 2006 Sep;111(3):855-76. doi: 10.1016/j.pharmthera.2006.02.001. Epub 2006 Mar 20. PMID 16545872
- [Background] Mansergh G, Koblin BA, Colfax GN, McKirnan DJ, Flores SA, Hudson SM; Project MIX Study Team. Preefficacy use and sharing of antiretroviral medications to prevent sexually-transmitted HIV infection among US men who have sex with men. J Acquir Immune Defic Syndr. 2010 Oct;55(2):e14-6. doi: 10.1097/QAI.0b013e3181f27616. No abstract available. PMID 20859085
- [Background] Wilson DP, Prestage GP, Gray RT, Hoare A, McCann P, Down I, Guy RJ, Drummond F, Klausner JD, Donovan B, Kaldor JM. Chemoprophylaxis is likely to be acceptable and could mitigate syphilis epidemics among populations of gay men. Sex Transm Dis. 2011 Jul;38(7):573-9. doi: 10.1097/OLQ.0b013e31820e64fd. PMID 21343845
- [Background] Carballo-Dieguez A, Bauermeister J, Ventuneac A, Dolezal C, Mayer K. Why rectal douches may be acceptable rectal-microbicide delivery vehicles for men who have sex with men. Sex Transm Dis. 2010 Apr;37(4):228-33. doi: 10.1097/OLQ.0b013e3181bf9b2d. PMID 19959973
- [Background] Liu A, Vittinghoff E, Irvin R, et al. Sexual frequency and planning among at-risk MSM in the US: implications for daily vs. intermittent pre-exposure prophylaxis (PrEP). 6th IAS Conference on HIV Pathogenesis and Treatment. Abstract no. TUPE362 2011; Rome, Italy.
- [Background] McConnell J. A Proposed Lexicon of Intermittent PrEP Possibilities. In: Subcommittee CPR, ed2009.
- [Background] Santos GM, Emenyonu NI, Bajunirwe F, Rain Mocello A, Martin JN, Vittinghoff E, Bangsberg DR, Hahn JA. Self-reported alcohol abstinence associated with ART initiation among HIV-infected persons in rural Uganda. Drug Alcohol Depend. 2014 Jan 1;134:151-157. doi: 10.1016/j.drugalcdep.2013.09.025. Epub 2013 Oct 5. PMID 24169501
- [Background] Hahn JA, Bwana MB, Javors MA, Martin JN, Emenyonu NI, Bangsberg DR. Biomarker testing to estimate under-reported heavy alcohol consumption by persons with HIV initiating ART in Uganda. AIDS Behav. 2010 Dec;14(6):1265-8. doi: 10.1007/s10461-010-9768-y. PMID 20697796
- [Background] Hahn JA, Fatch R, Kabami J, Mayanja B, Emenyonu NI, Martin J, Bangsberg DR. Self-Report of Alcohol Use Increases When Specimens for Alcohol Biomarkers Are Collected in Persons With HIV in Uganda. J Acquir Immune Defic Syndr. 2012 Dec 1;61(4):e63-4. doi: 10.1097/QAI.0b013e318267c0f1. No abstract available. PMID 23138732
- [Background] Armstrong AW, Watson AJ, Makredes M, Frangos JE, Kimball AB, Kvedar JC. Text-message reminders to improve sunscreen use: a randomized, controlled trial using electronic monitoring. Arch Dermatol. 2009 Nov;145(11):1230-6. doi: 10.1001/archdermatol.2009.269. PMID 19917951
- [Background] Cocosila M, Archer N, Haynes RB, Yuan Y. Can wireless text messaging improve adherence to preventive activities? Results of a randomised controlled trial. Int J Med Inform. 2009 Apr;78(4):230-8. doi: 10.1016/j.ijmedinf.2008.07.011. Epub 2008 Sep 7. PMID 18778967
- [Background] Franklin VL, Waller A, Pagliari C, Greene SA. A randomized controlled trial of Sweet Talk, a text-messaging system to support young people with diabetes. Diabet Med. 2006 Dec;23(12):1332-8. doi: 10.1111/j.1464-5491.2006.01989.x. PMID 17116184
- [Background] Granholm E, Ben-Zeev D, Link PC, Bradshaw KR, Holden JL. Mobile Assessment and Treatment for Schizophrenia (MATS): a pilot trial of an interactive text-messaging intervention for medication adherence, socialization, and auditory hallucinations. Schizophr Bull. 2012 May;38(3):414-25. doi: 10.1093/schbul/sbr155. Epub 2011 Nov 10. PMID 22080492
- [Background] Miloh T, Annunziato R, Arnon R, Warshaw J, Parkar S, Suchy FJ, Iyer K, Kerkar N. Improved adherence and outcomes for pediatric liver transplant recipients by using text messaging. Pediatrics. 2009 Nov;124(5):e844-50. doi: 10.1542/peds.2009-0415. Epub 2009 Oct 12. PMID 19822583
- [Background] Petrie KJ, Perry K, Broadbent E, Weinman J. A text message programme designed to modify patients' illness and treatment beliefs improves self-reported adherence to asthma preventer medication. Br J Health Psychol. 2012 Feb;17(1):74-84. doi: 10.1111/j.2044-8287.2011.02033.x. Epub 2011 Jun 22. PMID 22107110
- [Background] Rodgers A, Corbett T, Bramley D, Riddell T, Wills M, Lin RB, Jones M. Do u smoke after txt? Results of a randomised trial of smoking cessation using mobile phone text messaging. Tob Control. 2005 Aug;14(4):255-61. doi: 10.1136/tc.2005.011577. PMID 16046689
- [Background] Shapiro JR, Bauer S, Andrews E, Pisetsky E, Bulik-Sullivan B, Hamer RM, Bulik CM. Mobile therapy: Use of text-messaging in the treatment of bulimia nervosa. Int J Eat Disord. 2010 Sep;43(6):513-9. doi: 10.1002/eat.20744. PMID 19718672
- [Background] Wei J, Hollin I, Kachnowski S. A review of the use of mobile phone text messaging in clinical and healthy behaviour interventions. J Telemed Telecare. 2011;17(1):41-8. doi: 10.1258/jtt.2010.100322. Epub 2010 Nov 19. PMID 21097565
- [Background] Fuqua V, Chen YH, Packer T, Dowling T, Ick TO, Nguyen B, Colfax GN, Raymond HF. Using social networks to reach Black MSM for HIV testing and linkage to care. AIDS Behav. 2012 Feb;16(2):256-65. doi: 10.1007/s10461-011-9918-x. PMID 21390535

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via street outreach, recruitment flyers, sexual health clinics, needle exchanges, community organizations, bars, websites, and social media in San Francisco Bay Area.
Pre-assignment Details: Potential participants completed a brief telephone screen to assess initial eligibility and, if eligible, were scheduled for an in-person screening visit. All participants gave informed consent using University of California, San Francisco (UCSF) IRB-approved consent forms. Participants were evaluated for eligibility based on the inclusion criteria during the in-person screening visit.
Groups:
- Placebo: Placebo (identical capsule as treatment arm) 50mg, taken as needed
- Naltrexone: Naltrexone capsule, 50mg, taken as needed
Period: Overall Study
Arm/Group | Placebo | Naltrexone
Started | 60 | 60
Completed | 57 | 53
Not Completed | 3 | 7
Not completed — Lost to Follow-up | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo 50mg, as needed
  Placebo
- Naltrexone: Naltrexone 50mg, as needed
  Naltrexone
- Total: Total of all reporting groups
Arm/Group | Placebo | Naltrexone | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34 [30 to 42] | 38 [30 to 50] | 37 [30 to 45]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender Identity: Cis-gender male | 59 | 60 | 119
  Gender Identity: Transgender male (female to male) | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 32 | 33 | 65
  Asian | 4 | 2 | 6
  Black | 5 | 12 | 17
  Latino | 10 | 2 | 12
  Other | 9 | 11 | 20
Region of Enrollment [Count of Participants; unit: Participants] — All participants were from the San Francisco Bay Area.
  Participants
    United States | 60 | 60 | 120
Education [Count of Participants; unit: Participants]
  high school or less | 6 | 7 | 13
  some college | 19 | 17 | 36
  college or above | 35 | 36 | 71
Income [Count of Participants; unit: Participants]
  under $20,000 | 13 | 16 | 29
  $20 - 39,999 | 17 | 12 | 29
  $40,000 and above | 30 | 32 | 62
Employment [Count of Participants; unit: Participants]
  not employed | 14 | 21 | 35
  full-time | 29 | 28 | 57
  part-time | 12 | 9 | 21
  employed student | 5 | 2 | 7
Ever hospitalized for alcohol problem [Count of Participants; unit: Participants]
  No | 54 | 50 | 104
  Yes | 6 | 10 | 16
Ever received alcohol treatment [Count of Participants; unit: Participants]
  No | 43 | 42 | 85
  Yes | 8 | 11 | 19
  Missing | 9 | 7 | 16
Alcohol Craving Scale-Visual Analog [Median (Inter-Quartile Range); unit: units on a scale] — The Visual Analog Scale for Craving Alcohol measures the amount of alcohol craving that the participant experienced over the past 24 hours from 0 (not at all) to 100 (strongest ever). The higher score indicates a worse outcome.
  units on a scale | 25 [10 to 40] | 30 [10 to 50] | 30 [10 to 50]
HIV Status [Count of Participants; unit: Participants]
  HIV-positive | 17 | 14 | 31
  HIV-negative | 43 | 46 | 89
Has health insurance [Count of Participants; unit: Participants]
  No | 6 | 5 | 11
  Yes | 54 | 55 | 109
Has regular health care provider [Count of Participants; unit: Participants]
  No | 10 | 8 | 18
  Yes | 50 | 52 | 102
Center for Epidemiological Studies Depression scale (CES-D) [Median (Inter-Quartile Range); unit: units on a scale] — The Center for Epidemiological Studies Depression scale, known as CES-D, is a 20 question scale (Alpha >0.85) with total scores from 0 (min) to 60 (max) points. A score of 16 or more is considered that the participants are depressed and is a worse outcome.
  units on a scale | 13 [8 to 21] | 12 [7 to 20] | 12 [8 to 20]
Alcohol Use Disorder Identification Test (AUDIT) [Median (Inter-Quartile Range); unit: units on a scale] — The Alcohol Use Disorder Identification test or AUDIT-10 is a validated 10-item screening tool designed by the World Health Organization. The questions are scored from 0 to 4 points with a total ranging from 0 to 40 points. A participant with a total score of 8 to 14 points is considered to have a hazardous or harmful alcohol consumption. A participant with a total score of 15 points and above is considered to have a moderate to severe alcohol use disorder. The higher score indicates a worse outcome.
  units on a scale | 17 [14 to 22] | 16 [12 to 20] | 17 [13 to 22]

OUTCOME MEASURES:

1. Primary Outcome: Binge Drinking Days Per Week
Description: This outcome measure determines the mean number of binge drinking days among participants randomized to targeted naltrexone and placebo arms. The Center for Disease Control (CDC) defines binge drinking as consuming 5 or more drinks on an occasion for men or 4 or more drinks on an occasion for women.
Time Frame: 12 weeks
Population: The binge drinking days analysis between targeted naltrexone and placebo arms is different from the participant flow chart. The overall number of participants is calculated from those participants that completed the ACASI survey at week 12.
Measure: Mean (Standard Deviation); unit: days per week
Groups:
- Targeted Naltrexone/Placebo: Participants who were randomized to the Targeted Naltrexone and Placebo arms.
Arm/Group | Targeted Naltrexone/Placebo
Number analyzed (Participants) | 108
days per week
  Naltrexone Arm: number analyzed (Participants) | 54
  Naltrexone Arm | 1.056 (1.522)
  Placebo Arm: number analyzed (Participants) | 54
  Placebo Arm | 1.722 (1.698)

2. Primary Outcome: Positive Ethyl Glucuronide (EtG) Tests
Description: This outcome measure determines the number of participants with positive ethyl glucuronide tests among non-dependent MSM who were randomized to targeted naltrexone and placebo arms. Ethyl glucuronide (EtG) is a non-volatile, water-soluble, stable, direct metabolite of ethanol that can be detected in urine for 48 hours or sometimes 72 hours after drinking if there is heavy drinking.
Time Frame: 12 weeks
Population: A total of 50 participants were analyzed in the targeted naltrexone arm and 52 participants were analyzed in the placebo arm.
Measure: Count of Participants; unit: Participants
Groups:
- Targeted Naltrexone/Placebo: Participants randomized to targeted naltrexone or Placebo arms
Arm/Group | Targeted Naltrexone/Placebo
Number analyzed (Participants) | 102
Participants
  Targeted Naltrexone: number analyzed (Participants) | 50
  Targeted Naltrexone | 23
  Placebo: number analyzed (Participants) | 52
  Placebo | 29

3. Primary Outcome: Male Anal Sex Partners
Description: This outcome measure determines the mean number of male anal sex partners among non-dependent MSM randomized to targeted naltrexone and placebo arms.
Time Frame: 12 weeks
Population: The overall number of participants analyzed for Male anal sex partners is based on those who completed the week 12 ACASI survey. This is different than the participant flow. There were 54 participants in each arm of the study.
Measure: Mean (Standard Deviation); unit: sex partners
Groups:
- Targeted Naltrexone/Placebo: Participants randomized to targeted naltrexone (as needed) and placebo (as needed)
Arm/Group | Targeted Naltrexone/Placebo
Number analyzed (Participants) | 108
sex partners
  Targeted Naltrexone: number analyzed (Participants) | 54
  Targeted Naltrexone | 1.06 (1.41)
  Placebo: number analyzed (Participants) | 54
  Placebo | 1.98 (3.59)

4. Primary Outcome: Unprotected Anal Sex Partners While Intoxicated With Alcohol
Description: This outcome measure determines the mean number of unprotected anal sex partners while intoxicated with alcohol among targeted naltrexone and placebo arms .
Time Frame: 12 weeks
Population: The overall number of participants analyzed for Unprotected anal sex partners while intoxicated with alcohol is based on the number of participants who completed the week 12 survey. This is different than the participant flow. There were 54 participants in the targeted naltrexone and the placebo arms.
Measure: Mean (Standard Deviation); unit: partners
Groups:
- Targeted Naltrexone/Placebo: The participants in the targeted naltrexone (as needed) and placebo (as needed) arms
Arm/Group | Targeted Naltrexone/Placebo
Number analyzed (Participants) | 108
partners
  Targeted Naltrexone: number analyzed (Participants) | 54
  Targeted Naltrexone | 0.96 (1.52)
  Placebo: number analyzed (Participants) | 54
  Placebo | 0.56 (0.95)

5. Primary Outcome: HIV-serodiscordant Unprotected Anal Sex Partners
Description: This outcome measure determines the mean number of HIV-serodiscordant unprotected anal sex partners among the targeted naltrexone and placebo arms.
Time Frame: 12 weeks
Population: The overall number of participant analyzed for HIV-serodiscordant unprotected anal sex partners is based on the participants who completed the week 12 survey. This is different than the participant flow.
Measure: Mean (Standard Deviation); unit: partners
Groups:
- Targeted Naltrexone/Placebo: Participants that were randomized to targeted naltrexone (as needed) and placebo (as needed)
Arm/Group | Targeted Naltrexone/Placebo
Number analyzed (Participants) | 108
partners
  Targeted Naltrexone: number analyzed (Participants) | 54
  Targeted Naltrexone | 0.28 (0.45)
  Placebo: number analyzed (Participants) | 54
  Placebo | 0.26 (0.44)

6. Primary Outcome: Unprotected Anal Sex Events With Serodiscordant Partners
Description: This outcome measure determines the mean number of unprotected anal sex events with serodiscordant partners
Time Frame: 12 weeks
Population: The overall number of participants analyzed is based on those who completed the week 12 survey. This is different than the participant flow. There are 54 participants in each arm.
Measure: Mean (Standard Deviation); unit: events
Groups:
- Targeted Naltrexone/Placebo: Participants who were randomized to targeted naltrexone and placebo arms
Arm/Group | Targeted Naltrexone/Placebo
Number analyzed (Participants) | 108
events
  Targeted Naltrexone: number analyzed (Participants) | 54
  Targeted Naltrexone | 0.81 (2.0)
  Placebo: number analyzed (Participants) | 54
  Placebo | 0.41 (0.92)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Placebo | Naltrexone
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 1/60 | 1/60
Other Adverse Events (participants affected / at risk) | 20/60 | 43/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=60) | Naltrexone (N=60)
bowel obstructions (Gastrointestinal disorders) | 1 (1) | 0 (0)
soft-tissue infection (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=60) | Naltrexone (N=60)
nausea (Gastrointestinal disorders) | 4 (4) | 14 (14)
hyperglycemia (Renal and urinary disorders) | 9 (9) | 8 (8)
headache (Vascular disorders) | 2 (2) | 7 (7)
increased ALT (Hepatobiliary disorders) | 3 (3) | 5 (5)
increased AST (Hepatobiliary disorders) | 2 (2) | 6 (6)
rash (General disorders) | 0 (0) | 3 (3)
diarrhea (Metabolism and nutrition disorders) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
Future studies outside the San Francisco Bay Area and inclusive of other populations with mild to moderate AUD may be needed to examine the potential of targeted naltrexone more broadly. Our self-reported alcohol measures may be subject to bias. However, these measures have been validated and we have used ACASI to further enhance the validity of our self-reported measures. There is evidence that collecting alcohol biomarkers can enhance validity of self-report of alcohol use.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT02330419/Prot_SAP_000.pdf